CLINICAL TRIAL: NCT04183348
Title: Evaluation of the Effect of a Visio-Hearing Training Protocol on Spatial Hearing in Subjects With Hearing Loss
Acronym: EVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 69HCL19_0567
Record Dates: First submitted 2019-11-27; First posted 2019-12-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Cochlear Nerve Deafness; Cochlear Diseases; Cochlear Hearing Loss; Hearing Loss; Deafness
MeSH Terms: conditions — Retrocochlear Diseases; Cochlear Diseases; Hearing Loss, Sensorineural; Hearing Loss; Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): 10 normal hearing adults (NH) 10 unilateral deafness adults (SU) 10 mono-implanted adults (uIC) 10 bi-implanted adults (bIC)
  Interventions: Behavioral: Training Protocol n°1 first at Visit 1, then, Training Protocol n°2 at Visit 2
- Group B (Experimental): 10 normal hearing adults (NH) 10 unilateral deafness adults (SU) 10 mono-implanted adults (uIC) 10 bi-implanted adults (bIC)
  Interventions: Behavioral: Training Protocol n°2 first at Visit 1, then, Training Protocol n°1 at Visit 2

INTERVENTIONS:
Behavioral: Training Protocol n°1 first at Visit 1, then, Training Protocol n°2 at Visit 2 — During Protocol 1 (visit 1), participants of Group A will perform auditory spatial localization tasks with sensory feedback and during Protocol 2 (visit 2), they will perform auditory tasks without any notion of spatial localization. The 2 visits will be spaced at least 2 weeks (Wash-out).
  The effects of each of the protocols on spatial location hearing abilities will be specifically assessed by comparing the results of the different assessments (SPHERE and Visual Discrimination Test) obtained before and after each protocol.
  Arms: Group A
Behavioral: Training Protocol n°2 first at Visit 1, then, Training Protocol n°1 at Visit 2 — During Protocol 2 (visit 1), participants of Group B will perform auditory tasks without any notion of spatial localization and during Protocol 1 (visit 2), they will perform auditory spatial localization tasks with sensory feedback. The 2 visits will be spaced at least 2 weeks (Wash-out).
  The effects of each of the protocols on spatial location hearing abilities will be specifically assessed by comparing the results of the different assessments (SPHERE and Visual Discrimination Test) obtained before and after each protocol.
  Arms: Group B

SUMMARY:
We recently developed a new Neuro-immersion system based on virtual reality and 3D (dimension) motion tracking. This tool makes it possible to evaluate and record the spatial localization performance of sounds and to highlight localization deficits in the three dimensions of space in deaf patients. Unfortunately, there is currently no suitable support to compensate for these localization deficits. However, the discomfort felt by the patients is clearly verbalized.

Thanks to the new virtual reality system, we are now able to develop a training protocol based on spatial sound localization tasks.

ELIGIBILITY:
Inclusion Criteria:

For all participants (patients and normal hearing adults):

* Ages 18 and 65
* Normal vision (with or without correction)
* Able to understand experimental instructions
* Member of the social security scheme
* Informed of the study and signed the consent form

For hearing standards (NH):

- No hearing problems

For patients (SU, uIC and bIC):

* Regular follow-up in the ENT (Ear, nose, and throat) department of the Edouard Herriot Hospital in Lyon or the Purpan Hospital, in Toulouse
* Unilateral deep deafness (only for SU patients)
* Holder of one Cochlear implant for more than one year (only for uIC patients)
* Holder of the second Cochlear implant for more than one year (only for bIC patients)

Exclusion Criteria:

* Oculomotor disorder
* Bilateral vestibular areflexia
* Neurological and/or psychiatric history
* Person placed under legal protection, guardianship or trusteeship
* Pregnant or nursing woman

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Composite measure of spatial localization auditory tasks effect of each training protocol on spatial auditory performances | 1 day
  * Explicit spatial auditory performances ("2d-D") is the combined (head) pointing error, corresponding to the distance in the space between the exact position of the target and the pointing of the subject. In other words, the more precise the subject becomes in his location of a sound source and the lower the value of "2d-D".
  * Implicit spatial auditory performances (called "RT") is the response time between the participant's response and the light point.

SECONDARY OUTCOMES:
Measure of the sensory feedback effect on spatial auditory performance by comparing the composite measure of the two training protocols | 1 day
  * Explicit spatial auditory performances ("2d-D") is the combined (head) pointing error, corresponding to the distance in the space between the exact position of the target and the pointing of the subject. In other words, the more precise the subject becomes in his location of a sound source and the lower the value of "2d-D".
  * Implicit spatial auditory performances (called "RT") is the response time between the participant's response and the light point

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service d'Oto-Rhino-Laryngologie et Chirurgie cervico-faciale, Hôpital Edouard Herriot, Bron
  - Service d'Oto-Rhino-Laryngologie et Chirurgie cervico-faciale, Hôpital Purpan, CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valzolgher C, Bouzaid S, Grenouillet S, Gatel J, Ratenet L, Murenu F, Verdelet G, Salemme R, Gaveau V, Coudert A, Hermann R, Truy E, Farne A, Pavani F. Training spatial hearing in unilateral cochlear implant users through reaching to sounds in virtual reality. Eur Arch Otorhinolaryngol. 2023 Aug;280(8):3661-3672. doi: 10.1007/s00405-023-07886-1. Epub 2023 Mar 11. PMID 36905419